CLINICAL TRIAL: NCT00234429
Title: A Randomized, Placebo-Controlled, Double-Blind Phase 2b Study of Raltitrexed (Tomudex) and ZD1839 (Iressa) Versus Raltitrexed Alone as Second Line Chemotherapy in Subjects With Colorectal Carcinoma
Brief Title: A Phase 2 Study of Tomudex & Iressa as Second Line Chemotherapy in Subjects With Colorectal Carcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1839IL/0143
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Colorectal Cancer
Keywords: Colorectal carcinoma advanced disease
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Gefitinib; raltitrexed

INTERVENTIONS:
Drug: Gefitinib, raltitrexed

SUMMARY:
The primary objective of this study is to compare the activity of raltitrexed and ZD1839 versus raltitrexed alone as second line chemotherapy in subjects with colorectal carcinoma by estimating progression free survival (PFS) in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 75 years, inclusive
* histologically-confirmed metastatic colorectal carcinoma; measurable lesion according to the Response Evaluation Criteria in Solid Tumours (RECIST)
* relapsed after treatment with a fluoropyrimidine-based chemotherapy
* prior chemotherapeutic regimen for metastatic or locally advanced disease with an interval of at least 4 weeks between the last administration of chemotherapy an the first administration of study treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* life expectancy of at least 12 weeks

Exclusion Criteria:

* Known severe hypersensitivity to raltitrexed or any of the excipients of this product
* known severe hypersensitivity to raltitrexed or any of the excipients of this product
* active infection or uncontrolled diarrhoea
* cerebral metastasis or meningeal carcinomatosis
* any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded)
* simultaneous antitumoral treatment
* radiotherapy within 2 weeks before entry into the study
* other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* any unresolved chronic toxicity greater than common toxicity criteria (CTC) grade 2 from previous anticancer therapy (except alopecia)
* significant clinical disorder or laboratory finding (leukocyte count less than 3.0 x 109 /litre (L) or platelets less than 100 x 109 /L; serum total bilirubin more than 2.0 mg/dl; as judged by investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic, or renal disease); creatinine clearance ≥ 65ml/min (according to Cockcroft-Gault formula); alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2 times the upper limit of the reference range (ULRR) if no demonstrable liver metastases, or greater than 5 times the ULRR in the presence of liver metastases)
* pregnancy or breast feeding (women of child-bearing potential)
* concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or ST John's Wort;
* Treatment with a non- approved or investigational drug within 30 days before Day 1 of study treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74
Dates: Start 2003-11; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Determine the progression free survival

SECONDARY OUTCOMES:
Determine objective tumor response

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Spain Medical Director, MD, Study Director — AstraZeneca
Locations (9):
- Spain (9):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Gijón
  - Research Site, León
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Pamplona
  - Research Site, Valladolid

REFERENCES:
- [Derived] Zanni MV, Foldyna B, McCallum S, Burdo TH, Looby SE, Fitch KV, Fulda ES, Autissier P, Bloomfield GS, Malvestutto CD, Fichtenbaum CJ, Overton ET, Aberg JA, Erlandson KM, Campbell TB, Ellsworth GB, Sheth AN, Taiwo B, Currier JS, Hoffmann U, Lu MT, Douglas PS, Ribaudo HJ, Grinspoon SK. Sex Differences in Subclinical Atherosclerosis and Systemic Immune Activation/Inflammation Among People With Human Immunodeficiency Virus in the United States. Clin Infect Dis. 2023 Jan 13;76(2):323-334. doi: 10.1093/cid/ciac767. PMID 36101518
- [Derived] Looby SE, Kantor A, Burdo TH, Currier JS, Fichtenbaum CJ, Overton ET, Aberg JA, Malvestutto CD, Bloomfield GS, Erlandson KM, Cespedes M, Kallas EG, Masia M, Thornton AC, Smith MD, Flynn JM, Kileel EM, Fulda E, Fitch KV, Lu MT, Douglas PS, Grinspoon SK, Ribaudo HJ, Zanni MV. Factors Associated With Systemic Immune Activation Indices in a Global Primary Cardiovascular Disease Prevention Cohort of People With Human Immunodeficiency Virus on Antiretroviral Therapy. Clin Infect Dis. 2022 Oct 12;75(8):1324-1333. doi: 10.1093/cid/ciac166. PMID 35235653
- [Derived] Zanni MV, Currier JS, Kantor A, Smeaton L, Rivard C, Taron J, Burdo TH, Badal-Faesen S, Lalloo UG, Pinto JA, Samaneka W, Valencia J, Klingman K, Allston-Smith B, Cooper-Arnold K, Desvigne-Nickens P, Lu MT, Fitch KV, Hoffman U, Grinspoon SK, Douglas PS, Looby SE. Correlates and Timing of Reproductive Aging Transitions in a Global Cohort of Midlife Women With Human Immunodeficiency Virus: Insights From the REPRIEVE Trial. J Infect Dis. 2020 Jul 9;222(Suppl 1):S20-S30. doi: 10.1093/infdis/jiaa214. PMID 32645159